CLINICAL TRIAL: NCT01851564
Title: Effective Haemostasis Using Self-expandable Covered Mesh-metal Oesophageal Stents Versus Standard Endoscopic Therapy in the Treatment of Oesophageal Variceal Haemorrhage: A Multicentre, Open, Prospective, Randomised, Controlled Study.
Brief Title: RCT of Stent Versus Standard Therapy in Oesophageal Variceal Haemorrhage
Acronym: SOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Royal Free Hampstead NHS Trust (Other); Barts & The London NHS Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 74570; 11/0261 (Other: Sponsors Reference (UCL)); 13392 (Registry Identifier: UK Clinical Research Network Portfolio Database)
Record Dates: First submitted 2012-12-21; First posted 2013-05-10 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2015-06

CONDITIONS: Acute Bleeding Esophageal Varices
Keywords: Gastrointestinal Haemorrhage; Varices; Liver Cirrhosis; Stent
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Varicose Veins; Liver Cirrhosis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SEMS for primary variceal haemorrhage (Experimental): Use of the Self-expanding mesh-metal oesophageal stent (SEMS) as primary therapy for Acute Variceal Haemorrhage.
  Interventions: Device: Self-expanding mesh-metal oesophageal stent (SEMS)
- Standard Therapy - Primary Haemorrhage (Active Comparator): Use of standard medical and endoscopic therapy for the treatment of primary variceal haemorrhage.
  Interventions: Other: Standard Therapy
- SEMS for Failure to Control Bleeding (Experimental): Use of the self expanding mesh-metal stent for failure of standard therapy in oesophageal variceal haemorrhage.
  Interventions: Device: Self-expanding mesh-metal oesophageal stent (SEMS)
- Standard Therapy - Failure of Control (Active Comparator): Use of standard medical and endoscopic therapy for failure of standard therapy in oesophageal variceal haemorrhage.
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Device: Self-expanding mesh-metal oesophageal stent (SEMS) — A removable stent designed for the treatment of bleeding oesophageal varices.
  Other Names: DANIS Stent
  Arms: SEMS for Failure to Control Bleeding; SEMS for primary variceal haemorrhage
Other: Standard Therapy — Standard Medical and Endoscopic Therapy
  Arms: Standard Therapy - Failure of Control; Standard Therapy - Primary Haemorrhage

SUMMARY:
The mortality rates from Acute Variceal Haemorrhage remain significant and first line therapy may fail in 15-25% of patients. The self-expandable metal stent has been described in case series as having a very high efficacy at control of haemorrhage from oesophageal varices when used as rescue therapy. This randomised controlled trial aims to assess for any potential superiority of the stent over 'standard' endoscopic techniques as primary or rescue therapy for bleeding oesophageal varices.

DETAILED DESCRIPTION:
Despite improvements in recent years, mortality from variceal bleeding remains significant. The routine use of banding ligation, vasoactive drugs, and antibiotics has had an impact on survival rates such that survival rates of patients with Childs-Pugh A and B class cirrhosis may be as high as 90% at 30 days. However, the successful outcome of variceal bleeding is compromised in some patients because of initial failure to control bleeding or early re-bleeding, both of which have a significant impact on mortality.

The SX-Ella Danis stent (Ella-CS, Hradec Kralove, Czech Republic) is a removable, covered, self-expanding mesh-metal stent (SEMS) that can be deployed in the lower oesophagus over an endoscopically placed guidewire without radiological screening. The stent controls bleeding by tamponade of varices in the lower oesophagus.

The series reported to date suggest that the self-expandable covered stents can provide 100% haemostasis rates when applied for refractory oesophageal variceal bleeding. Given the potentially lower risks of re-bleeding and safe, easy insertion techniques the self-expandable covered stents may offer a superior alternative to standard endoscopic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Arm 1: Participants with Child-Pugh grade B or C cirrhosis with variceal haemorrhage, where the bleeding is from a site which would ordinarily be treated with band ligation . The diagnosis of cirrhosis may be proven by previous histology or suspected using clinical, radiological and biochemical data.
* Arm 2: Participants with Child-Pugh grade A, B or C cirrhosis who present with failure to control bleeding within 5 days of an initial attempt at standard endoscopic therapy of acute haemorrhage from a site which would ordinarily be treated with band ligation.

Exclusion Criteria:

* < 18 Years of age
* Child-Pugh grade A cirrhosis (for Arm 1 only)
* Varices which would not be treated with band ligation as standard therapy
* Non-cirrhotic portal hypertension
* Malignancy of the oesophagus, stomach or upper respiratory tract
* Oesophageal stenosis which prohibits endoscopy
* Recent oesophageal surgery
* A large hiatus hernia which prevents stent placement
* Known hepatocellular carcinoma considered to be incurable (according to Milan Criteria)
* Patients in the terminal phases of hepatological or other disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-08; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Failure to Control Bleeding | 7 days
  Failure to control Bleeding (as defined by the Baveno V Criteria) or re-bleeding within 7 days.

SECONDARY OUTCOMES:
Absence of Bleeding at 14 and 42 days | 14 and 42 days
Participant Survival | 7, 14, 42 days and 6 months
Absence of Stent Migration | 7 days
  for the duration of stent migration
Requirement for Blood products | 7 days
Requirement for Analgesia and Sedation whilst Stent in in situ | 7 days
Presence of Thoracic Pain or Dysphagia | 7 days
Length of Intensive Care Unit and Total Hospital Stay | Total Length of Intensive Care Unit and Hospital Stay (an average of 3 and 10 days respectively)
Requirement for additional endoscopic therapy or salvage therapy (such as TIPS) | 7 days
Repeated presentation with variceal bleeding within 6 months | 6 months

OTHER OUTCOMES:
Unexpected Serious Adverse Device Effect | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: James O'Beirne, MBBS FRCP, Principal Investigator — Royal Free London NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - United Bristol Hospitals NHS Foundation Trust, Bristol
  - Barts Health NHS Trust, London
  - Royal Free London NHS Foundation Trust, London

REFERENCES:
- [Background] Carbonell N, Pauwels A, Serfaty L, Fourdan O, Levy VG, Poupon R. Improved survival after variceal bleeding in patients with cirrhosis over the past two decades. Hepatology. 2004 Sep;40(3):652-9. doi: 10.1002/hep.20339. PMID 15349904
- [Background] Burroughs AK, Triantos CK, O'Beirne J, Patch D. Predictors of early rebleeding and mortality after acute variceal hemorrhage in patients with cirrhosis. Nat Clin Pract Gastroenterol Hepatol. 2009 Feb;6(2):72-3. doi: 10.1038/ncpgasthep1336. Epub 2008 Dec 17. PMID 19092789
- [Background] Ben-Ari Z, Cardin F, McCormick AP, Wannamethee G, Burroughs AK. A predictive model for failure to control bleeding during acute variceal haemorrhage. J Hepatol. 1999 Sep;31(3):443-50. doi: 10.1016/s0168-8278(99)80035-x. PMID 10488702
- [Background] D'Amico G, De Franchis R; Cooperative Study Group. Upper digestive bleeding in cirrhosis. Post-therapeutic outcome and prognostic indicators. Hepatology. 2003 Sep;38(3):599-612. doi: 10.1053/jhep.2003.50385. PMID 12939586
- [Background] de Franchis R; Baveno V Faculty. Revising consensus in portal hypertension: report of the Baveno V consensus workshop on methodology of diagnosis and therapy in portal hypertension. J Hepatol. 2010 Oct;53(4):762-8. doi: 10.1016/j.jhep.2010.06.004. Epub 2010 Jun 27. No abstract available. PMID 20638742
- [Background] Hubmann R, Bodlaj G, Czompo M, Benko L, Pichler P, Al-Kathib S, Kiblbock P, Shamyieh A, Biesenbach G. The use of self-expanding metal stents to treat acute esophageal variceal bleeding. Endoscopy. 2006 Sep;38(9):896-901. doi: 10.1055/s-2006-944662. PMID 16981106
- [Background] Zehetner J, Shamiyeh A, Wayand W, Hubmann R. Results of a new method to stop acute bleeding from esophageal varices: implantation of a self-expanding stent. Surg Endosc. 2008 Oct;22(10):2149-52. doi: 10.1007/s00464-008-0009-7. Epub 2008 Jul 12. PMID 18622540
- [Background] Wright G, Lewis H, Hogan B, Burroughs A, Patch D, O'Beirne J. A self-expanding metal stent for complicated variceal hemorrhage: experience at a single center. Gastrointest Endosc. 2010 Jan;71(1):71-8. doi: 10.1016/j.gie.2009.07.028. Epub 2009 Oct 30. PMID 19879564
- [Background] Sarin SK, Kumar A. Gastric varices: profile, classification, and management. Am J Gastroenterol. 1989 Oct;84(10):1244-9. PMID 2679046
- [Background] Garcia-Tsao G, Sanyal AJ, Grace ND, Carey W; Practice Guidelines Committee of the American Association for the Study of Liver Diseases; Practice Parameters Committee of the American College of Gastroenterology. Prevention and management of gastroesophageal varices and variceal hemorrhage in cirrhosis. Hepatology. 2007 Sep;46(3):922-38. doi: 10.1002/hep.21907. No abstract available. PMID 17879356